CLINICAL TRIAL: NCT03176875
Title: Comparison of Partial and Exclusive Enteral Nutrition in the Treatment of Active Childhood-onset Crohn's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Darja Urlep, Principal investigator, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20150146
Record Dates: First submitted 2017-05-25; First posted 2017-06-06 (Actual); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: Adolescent; Child; Diet; Crohn Disease; Enteral Nutrition; Remission
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEN group (Experimental): Partial enteral nutrition (PEN) group will receive 75% of their daily dietary needs from a polymeric formula (Alicalm, Nutricia) and a limited (25% of dietary needs = 1 meal per day) from an antiinflammatory diet for CD (AID-CD) for 6 weeks.
  Interventions: Other: ALICALM (75% of daily caloric requirements)
- EEN group (Active Comparator): Exclusive enteral nutrition (EEN) group will receive 100 % of their daily caloric requirements from a poymeric formula (Alicalm, Nutricia) for 6 weeks.
  Interventions: Other: ALICALM (100% of daily caloric requirements)

INTERVENTIONS:
Other: ALICALM (75% of daily caloric requirements) — PEN group will receive 75% of their daily dietary needs from a polymeric formula (Alicalm, Nutricia) and 25% of daily dietary needs (1 meal per day) from an antiinflammatory diet for CD (AID-CD) for 6 weeks.
  Arms: PEN group
Other: ALICALM (100% of daily caloric requirements) — EEN group will receive 100% of their daily dietary needs from a polymeric formula (Alicalm, Nutricia) for 6 weeks.
  Arms: EEN group

SUMMARY:
The primary objective of this study is to determine the efficacy of a novel enteral nutrition (EN) protocol (delivering 75% of patient's caloric needs through EN) for induction of remission in patients with active childhood-onset Crohn's disease (CD) and compare it to the standard protocol with exclusive enteral nutrition (EEN). This novel approach allows patients to consume remaining calories (25%) from an antiinflammatory diet for CD (AID-CD).

The hypothesis is that no significant difference in the remission rate between the novel EN protocol with partial enteral nutrition (PEN) and standard protocol with EEN will be observed.

DETAILED DESCRIPTION:
Background: Exclusive enteral nutrition (EEN) is a well established method of treatment for inducing remission in childhood-onset Crohn's disease. It involves placing children on a strict diet composed only of a single polymeric formula, as the sole source of nutrition over 6 to 8 weeks. Use of this treatment method results in clinical remission in 50% to 80% of children by week 6-8.

Partial enteral nutrition (PEN) would be more acceptable to patients than EEN, and might be an effective treatment for active Crohn's disease. Moreover, there are studies suggesting that PEN may be effective for the induction of remission in pediatric patients with Crohn's disease; however, the level of evidence is still low.

Methods: This is a prospective randomized controlled trial, in patients with active childhood-onset Crohn's disease comparing two arms over 6 weeks of therapy.

Group 1 (PEN group): will receive 75% of their dietary needs from a polymeric formula (Alicalm, Nutricia) and a limited (25% of dietary needs = 1 meal per day) whole food AID-CD for 6 weeks.

Group 2 (EEN group): will receive EEN with Alicalm (Nutricia) for 6 weeks.

Patients will be seen at onset and week 1, 3, and 6.

This study will evaluate clinical response (a decrease in PCDAI score of ≥12.5 points), clinical remission (PCDAI <10) and mucosal healing using SES-CD in both groups, as well as the effects of the two nutritional approaches on the patients' nutritional status.

Antiinflammatory diet for Crohn's disease (AID-CD) is based on reducing exposure to animal fat, simple carbohydrates and processed food. We removed foods that previous research has shown to induce inflammation and added foods that have been shown to be beneficial in reducing inflammation. Our AID-CD is based on Central European and thus Slovenian local and traditional cuisine.

ELIGIBILITY:
Inclusion Criteria:

* Children (4 - 18 years of age)
* Young adults (>18 and ≤ 30 years of age) with childhood-onset CD (the diagnosis of CD before 18 years of age)
* Assured diagnosis of Crohn's disease according to the Porto criteria
* Patients with Active CD (Pediatric Crohn's Disease Activity Index (PCDAI) ≥10 in children or Harvey-Bradshaw Index (HBI) >3 in young adults )
* Patients with new-onset CD and patients with active disease despite stable doses of concomitant therapy with immunomodulators (thiopurines, methotrexate, tacrolimus) for ≥ 3 months, on stable doses of biologic therapy (anti-TNF-a agents) for ≥ 2 months
* Patients will not be excluded if they start therapy with thiopurine concurrently, as thiopurines are not considered sufficient to induce remission in active disease before 8 weeks
* Written consent of the patient and/or the legal guardian

Exclusion Criteria:

* Patients with no disease activity ( PCDAI <10)
* Patients who have received corticosteroids of any kind in the previous 4 weeks.
* Patients with penetrating disease (abscess or fistula)
* Active Perianal disease
* Active Extraintestinal disease
* Sclerosing Cholangitis
* Patients with fixed stricture or small bowel obstruction
* If the patients had received any other medication for inducing remission such as steroids and/or antibiotics
* No consent of the patient and/or the legal guardian

Ages: 4 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-05-25 (Actual); Primary Completion 2018-07-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical Remission | 6 weeks
  Clinical Remission (Pediatric Crohn's Disease Activity Index <10) on an intention to treat principle after 6 weeks of therapy.

SECONDARY OUTCOMES:
Clinical response | 6 weeks
  - Clinical response defined as a decrease in Pediatric Crohn's Disease Activity Index score of ≥12.5 points) for children or a drop in HBI of at least 2 points in young adults
Mucosal healing | 6-8 weeks
  Mucosal healing using the Simple Endoscopic Score for CD (SES-CD)
Change in SES-CD | At week 0 and 6 -8 weeks following enrollment
  Change in SES-CD from baseline to 6 weeks
Changes in specific blood tests | At the 1, 3 and 6 weeks visits
  Changes in specific blood tests such as erythrocyte sedimentation rate (ESR), C reactive protein, hemoglobin, albumin, and platelets from baseline to 6 weeks
Changes in stool calprotectin concentrations | At the 3 and 6 weeks visits
  Changes in stool calprotectin concentrations (mg/kg) from baseline to 6 weeks
Changes in weight-z-scores | At the 0 and 6 weeks visits
  Changes in weight-z-scores
Changes in ITM -z-scores | At the 0 and 6 weeks visits
  Changes in ITM -z-scores

CONTACTS AND LOCATIONS:
Overall Officials: Rok Orel, MD, PhD, Study Chair — University Medical Centre Ljubljana, University Children's Hospital Ljubljana, Department of gastroenterology, hepatology and nutrition
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gupta K, Noble A, Kachelries KE, Albenberg L, Kelsen JR, Grossman AB, Baldassano RN. A novel enteral nutrition protocol for the treatment of pediatric Crohn's disease. Inflamm Bowel Dis. 2013 Jun;19(7):1374-8. doi: 10.1097/MIB.0b013e318281321b. PMID 23567777
- [Background] Sigall-Boneh R, Pfeffer-Gik T, Segal I, Zangen T, Boaz M, Levine A. Partial enteral nutrition with a Crohn's disease exclusion diet is effective for induction of remission in children and young adults with Crohn's disease. Inflamm Bowel Dis. 2014 Aug;20(8):1353-60. doi: 10.1097/MIB.0000000000000110. PMID 24983973
- [Derived] Urlep D, Benedik E, Brecelj J, Orel R. Partial enteral nutrition induces clinical and endoscopic remission in active pediatric Crohn's disease: results of a prospective cohort study. Eur J Pediatr. 2020 Mar;179(3):431-438. doi: 10.1007/s00431-019-03520-7. Epub 2019 Nov 28. PMID 31781933